CLINICAL TRIAL: NCT01072396
Title: A Randomized, Double-blind, Placebo-controlled, 6-week, Crossover Study to Examine the Effects of Tiotropium (Spiriva® HandiHaler®, 18 µg Once Daily) on Dynamic Hyperinflation and Physical Exercise Capacity in Patients With Early Stage Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Effects of Tiotropium on Breathing Capacity and Exercise Limitation in Early Stages of Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 205.440
Record Dates: First submitted 2010-02-19; First posted 2010-02-22 (Estimated); Results first posted 2013-05-15 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-04

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide

ARMS (3):
- 18 mcg tiotropium (Active Comparator): Patient to receive 1 tiotropium bromide inhalation powder capsule daily (in the morning) via HandiHaler
  Interventions: Drug: Tiotropium
- Placebo (Placebo Comparator): Patient to receive 1 placebo inhalation powder capsule daily (in the morning) identical to those containing tiotropium bromide inhalation powder via HandiHaler
  Interventions: Drug: Placebo
- Control (No Intervention): Age and gender matched control subjects to conduct incremental and constant work rate exercise tests for comparison to subjects with early stage COPD

INTERVENTIONS:
Drug: Tiotropium — double blind randomized crossover
  Arms: 18 mcg tiotropium
Drug: Placebo — inhalation powder capsule identical to those containing tiotropium bromide inhalation powder
  Arms: Placebo

SUMMARY:
Optimal clinical management in early stages of COPD is not established. Tiotropium has been shown to improve exercise tolerance during (CWR) cycle ergometry with GOLD stage II to IV COPD, improvements in constant speed treadmill time in a study of patients who also received pulmonary rehabilitation in a population of patients with predominantly severe and very severe disease (GOLD stages III and IV) and improvements in exertional dyspnea, and Shuttle Walk Test distance in GOLD stage III and IV COPD. However, data are lacking on the benefits of tiotropium on exercise tolerance in a patients with early stages of COPD who are symptomatic. Patients with milder ventilatory limitations (GOLD stages I/II COPD patients) may benefit from maintenance therapy and there is limited data on exercise limitation in patients with early stage COPD who are symptomatic. This study is designed to evaluate the mechanisms of breathlessness and assess physical activity limitation in early stage COPD patients compared to age and gender matched controls and will secondly investigate the effectiveness of treatment with tiotropium in improving dyspnea during exercise and exercise duration as a result of the bronchodilation effects of tiotropium leading to a reduction of dynamic hyperinflation in Early Stage COPD patients.

ELIGIBILITY:
Inclusion criteria:

For COPD subjects: Male or female, age of 40 years or older, smoking history >10 pack-years, symptomatic defined as baseline dyspnea index focal score of 9 or more and / or daily cough with production of sputum for three months per year during at least two consecutive years, diagnosis of early stage COPD according to: post-bronchodilator FEV1/FVC ratio <70%., FEV1 >/=50% post-bronchodilator predicted normal, and a decreased Inspiratory Capacity during exercise. For Age / Gender Matched Controls: Male or female, age of 40 years or older, nonsmoker, with no significant diseases.

Exclusion criteria:

Patients with a significant disease other than COPD; a significant disease is defined as a disease which, in the opinion of the investigator, may (i) put the patient at risk because of participation in the study, (ii) influence the results of the study, or (iii) cause concern regarding the patient's ability to participate in the study.

Patients with a history of asthma, Patients requiring the use of supplemental oxygen therapy, Patients who have a limitation of exercise performance as a result of factors other than fatigue or exertional dyspnoea, such as arthritis in the leg, angina pectoris, claudication or other conditions, or Patients with contraindications to exercise.

Note: Additional exclusion criteria for Age / Gender Matched Controls: Patients with a significant disease including COPD.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2010-02; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (15):
- United States (11):
  - 205.440.1006 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 205.440.1015 Boehringer Ingelheim Investigational Site, Jasper, Alabama
  - 205.440.1002 Boehringer Ingelheim Investigational Site, Torrance, California
  - 205.440.1018 Boehringer Ingelheim Investigational Site, Hartford, Connecticut
  - 205.440.1008 Boehringer Ingelheim Investigational Site, Springfield, Illinois
  - 205.440.1017 Boehringer Ingelheim Investigational Site, Muncie, Indiana
  - 205.440.1020 Boehringer Ingelheim Investigational Site, Livonia, Michigan
  - 205.440.1011 Boehringer Ingelheim Investigational Site, Lebanon, New Hampshire
  - 205.440.1019 Boehringer Ingelheim Investigational Site, Charlotte, North Carolina
  - 205.440.1013 Boehringer Ingelheim Investigational Site, Pittsburgh, Pennsylvania
  - 205.440.1007 Boehringer Ingelheim Investigational Site, Spartanburg, South Carolina
- Canada (4):
  - 205.440.2003 Boehringer Ingelheim Investigational Site, Kingston, Ontario
  - 205.440.2001 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 205.440.2004 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 205.440.2002 Boehringer Ingelheim Investigational Site, Ste-Foy, Quebec

REFERENCES:
- [Derived] Porszasz J, Blonshine S, Cao R, Paden HA, Casaburi R, Rossiter HB. Biological quality control for cardiopulmonary exercise testing in multicenter clinical trials. BMC Pulm Med. 2016 Jan 16;16:13. doi: 10.1186/s12890-016-0174-8. PMID 26775292
- [Derived] Gagnon P, Casaburi R, Saey D, Porszasz J, Provencher S, Milot J, Bourbeau J, O'Donnell DE, Maltais F. Cluster Analysis in Patients with GOLD 1 Chronic Obstructive Pulmonary Disease. PLoS One. 2015 Apr 23;10(4):e0123626. doi: 10.1371/journal.pone.0123626. eCollection 2015. PMID 25906326
- [Derived] Casaburi R, Maltais F, Porszasz J, Albers F, Deng Q, Iqbal A, Paden HA, O'Donnell DE; 205.440 Investigators. Effects of tiotropium on hyperinflation and treadmill exercise tolerance in mild to moderate chronic obstructive pulmonary disease. Ann Am Thorac Soc. 2014 Nov;11(9):1351-61. doi: 10.1513/AnnalsATS.201404-174OC. PMID 25289942
- [Derived] O'Donnell DE, Maltais F, Porszasz J, Webb KA, Albers FC, Deng Q, Iqbal A, Paden HA, Casaburi R; 205.440 investigators. The continuum of physiological impairment during treadmill walking in patients with mild-to-moderate COPD: patient characterization phase of a randomized clinical trial. PLoS One. 2014 May 1;9(5):e96574. doi: 10.1371/journal.pone.0096574. eCollection 2014. PMID 24788342

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study has two stages, in the first (exploratory) stage, the Control group (Healthy volunteer) is compared to the age-gender matched COPD patients in terms of baseline characteristics. In the second (confirmatory) stage, Placebo and Tiotropium are compared using a cross-over. Since the first stage is exploratory it is not reported.
Groups:
- Placebo/Tiotropium: Patients were randomized to receive treatment with Placebo for six weeks followed by treatment with Tiotropium 18 micrograms for six weeks
- Tiotropium/Placebo: Patients were randomized to receive treatment with Tiotropium 18 micrograms for six weeks followed by treatment with placebo for six weeks
Period: Period One
Arm/Group | Placebo/Tiotropium | Tiotropium/Placebo
Started | 63 | 63
Completed | 58 | 61
Not Completed | 5 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Protocol Violation | 2 | 1
Not completed — Withdrawal by Subject | 2 | 0
Period: Washout Period
Arm/Group | Placebo/Tiotropium | Tiotropium/Placebo
Started | 58 | 61
Completed | 58 | 60
Not Completed | 0 | 1
Not completed — Missing termination information | 0 | 1
Period: Period Two
Arm/Group | Placebo/Tiotropium | Tiotropium/Placebo
Started | 58 | 60
Completed | 57 | 57
Not Completed | 1 | 3
Not completed — Adverse Event | 0 | 3
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/Tiotropium | Tiotropium/Placebo | Total
Number analyzed (Participants) | 63 | 63 | 126
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (9.1) | 60.5 (8.6) | 61.2 (8.8)
Age, Customized [Number; unit: Participants]
  <=55 years | 14 | 21 | 35
  >55 to <=65 years | 28 | 23 | 51
  >65 years | 21 | 19 | 40
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 33 | 61
  Male | 35 | 30 | 65
Race/Ethnicity, Customized [Number; unit: Participants]
  Black | 6 | 6 | 12
  White | 57 | 57 | 114
Smoking Status [Number; unit: Participants]
  Ex-smoker | 33 | 34 | 67
  Currently smokes | 30 | 29 | 59
Smoking history [Mean (Standard Deviation); unit: pack years] | 46.0 (24.4) | 48.1 (20.0) | 47.0 (22.3)
Duration of COPD (Chronic Obstructive Pulmonary Disease) [Mean (Standard Deviation); unit: years] | 4.4 (4.6) | 5.3 (5.7) | 4.9 (5.2)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Inspiratory Capacity (IC) at Isotime
Description: Inspiratory capacity (IC) during CWR exercise testing measured at isotime (isotime was established during CWR exercise testing at baseline). Isotime is the minimum exercise time among all tests. Constant work rate exercise means the exercise is done under constant work rate.
Time Frame: baseline, six weeks of treatment
Population: Full Analysis Set (FAS) includes all patients with at least one baseline (at Visit 3 or 5) and two non-missing post-dosing data (at Visits 4 and 6) for the primary endpoint.
Measure: Least Squares Mean (Standard Error); unit: liter
Groups:
- Placebo: Patients who received placebo in period one or period two
- Tiotropium: Patients who received tiotropium in period one or period two
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 111 | 111
liter | 0.0035 (0.02) | 0.07 (0.02)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Placebo versus Tiotropium - crossover design; Test type: Superiority or Other; p = 0.0087, Mixed Models Analysis — Based on mixed effect model with repeated measures (MMRM) with fixed categorical effects for treatment, period and random effect for patient. Period baseline and patient baseline (average of two period baselines) were covariates in the model; Restricted maximum likelihood (REML) based MMRM; Mean Difference (Final Values) = 0.06, 95% CI [0.02 to 0.11]

2. Secondary Outcome: Constant Work Rate (CWR) Endurance Time
Description: CWR exercise duration calculated as the length of time of the exercise period
Time Frame: six weeks of treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 111 | 111
seconds | 6.0796 (0.0313) | 6.1458 (0.0313)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Placebo versus Tiotropium - corssover design; Test type: Superiority or Other; p = 0.0670, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Restricted maximum likelihood (REML) based MMRM; Adjusted mean ratio = 1.0685, 95% CI [0.9953 to 1.1470]

3. Secondary Outcome: Change From Baseline in Modified Borg Scale Ratings for Dyspnea Intensity at Isotime
Description: Modified Borg Scale is a participant rating of the intensity of dyspnea measured on a scale ranging from 0 (Nothing at all) to 10 (Maximal, most severe ever experienced).
Time Frame: baseline, six weeks of treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 111 | 111
Scores on a scale | -0.0485 (0.1330) | -0.2544 (0.1330)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Placebo versus Tiotropium - corssover design; Test type: Superiority or Other; p = 0.2417, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Restricted maximum likelihood (REML) based MMRM; Mean Difference (Final Values) = -0.2059, 95% CI [-0.5527 to 0.1408]

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Placebo | Tiotropium
Serious Adverse Events (participants affected / at risk) | 2/123 | 1/121
Other Adverse Events (participants affected / at risk) | 0/123 | 0/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=123) | Tiotropium (N=121)
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lentigo maligna stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.